CLINICAL TRIAL: NCT02036502
Title: A Phase I Multi-Cohort Trial of Pembrolizumab (MK-3475) in Combination With Backbone Treatments for Subjects With Multiple Myeloma
Brief Title: A Study of Pembrolizumab (MK-3475) in Combination With Standard of Care Treatments in Participants With Multiple Myeloma (MK-3475-023/KEYNOTE-023)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-023; 2013-003512-44 (EudraCT Number); MK-3475-023 (Other: Merck); KEYNOTE-023 (Other: Merck)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Multiple Myeloma
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab; Lenalidomide; Dexamethasone; Calcium Dobesilate; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1:pembro 2mg/kg+len 25mg+dex 40 mg (Experimental): Participants in Part 1 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 2 mg/kg once every 2 weeks (Q2W) (Days 1 and 15) in combination with lenalidomide 25 mg (Days 1-21) and dexamethasone 40 mg once weekly (Q1W) during Cycle 1 (28-day cycle).
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone
- Part 1:pembro 2mg/kg+len 10 mg+dex 40 mg (Experimental): Participants in Part 1 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 2 mg/kg Q2W (Days 1 and 15) in combination with lenalidomide 10 mg (Days 1-21) and dexamethasone 40 mg Q1W during Cycle 1 (28-day cycle).
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone
- Part 2:pembro 200 mg+len 25 mg+dex 40 mg (Experimental): Participants in Part 2 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 200 mg Q2W (Days 1 and 15) in combination with lenalidomide 25 mg (Days 1-21) and dexamethasone 40 mg Q1W during Cycle 1 (28-day cycle).
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone
- Part 2:pembro 200 mg+len 25 mg+dex 20 mg (Experimental): Participants in Part 2 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 200 mg Q2W (Days 1 and 15) in combination with lenalidomide 25 mg (Days 1-21) and dexamethasone 20 mg Q1W during Cycle 1 (28- day cycle).
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone
- Part 2:pembro 200 mg+len 10 mg+dex 40 mg (Experimental): Participants in Part 2 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 200 mg Q2W (Days 1 and 15) in combination with lenalidomide 10 mg (Days 1-21) and dexamethasone 40 mg Q1W during Cycle 1 (28-day cycle).
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone
- Part 3:pembro 200 mg+len 25 mg+dex 40 mg (Experimental): Participants in Part 3 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 200 mg Q2W (Days 1 and 15) in combination with lenalidomide 25 mg (Days 1-21) and dexamethasone 40 mg Q1W weekly during each 28-day cycle.
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone
- Part 3:pembro 200 mg+len 25 mg+dex 20 mg (Experimental): Participants in Part 3 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 200 mg Q2W (Days 1 and 15) in combination with lenalidomide 25 mg (Days 1-21) and dexamethasone 20 mg Q1W weekly during each 28-day cycle.
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone
- Part 3:pembro 200 mg+carf 56 mg/m^2+dex 20 mg (Experimental): Participants in Part 3 with relapsed or refractory multiple myeloma (rMM) received pembrolizumab 200 mg Q3W in combination with carfilzomib 56 mg/m^2 (Days 1, 2, 8, 9, 15, 16) and dexamethasone 20 mg once or twice weekly (Days 1, 2, 8, 9, 15, 16, 22, 23) during each 28-day cycle.
  Interventions: Biological: Pembrolizumab; Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous (IV) infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenalidomide — Oral capsule
  Other Names: REVLIMID®
  Arms: Part 1:pembro 2mg/kg+len 10 mg+dex 40 mg; Part 1:pembro 2mg/kg+len 25mg+dex 40 mg; Part 2:pembro 200 mg+len 10 mg+dex 40 mg; Part 2:pembro 200 mg+len 25 mg+dex 20 mg; Part 2:pembro 200 mg+len 25 mg+dex 40 mg; Part 3:pembro 200 mg+len 25 mg+dex 20 mg; Part 3:pembro 200 mg+len 25 mg+dex 40 mg
Drug: Dexamethasone — Oral tablet IV infusion
  Other Names: DECADRON®
Drug: Carfilzomib — IV infusion
  Other Names: KYPROLIS®
  Arms: Part 3:pembro 200 mg+carf 56 mg/m^2+dex 20 mg

SUMMARY:
This is a study of pembrolizumab (MK-3475) in combination with lenalidomide and low-dose dexamethasone in participants with refractory or relapsed and refractory Multiple Myeloma (rrMM), and in combination with carfilzomib and low-dose dexamethasone in participants with relapsed or refractory Multiple Myeloma (rMM).

This study was being done to find the maximum tolerated dose (MTD)/maximum administered dose (MAD) and recommended Phase 2 dose (RP2D), and to evaluate the safety and tolerability of pembrolizumab when given in combination with standard of care (SOC) treatments in participants with rrMM or rMM. Preliminary efficacy data will also be assessed. There was no primary hypothesis associated with this study.

On 03-Jul-2017, the United States Food and Drug Administration (US FDA) placed the rrMM cohort of this protocol on clinical hold based on safety data from two other pembrolizumab protocols: MK-3475-183 (NCT02576977) and MK-3475-185 (NCT02579863) presented to the Data Monitoring Committee.

On 15-Sep-2017, the US FDA placed the rMM cohort of this study on partial clinical hold. Enrollment was stopped and will not be reopened. Participants who are deriving clinical benefit were allowed to continue receiving study treatment until protocol-specific end of treatment, and then progress into long term safety and survival follow up. Participants who are not deriving clinical benefit, must stop study treatment and move into the long term safety and survival follow up.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Confirmed diagnosis of multiple myeloma (MM)
* MM with measurable disease
* Archival or newly obtained bone marrow material available. In addition, for participants in the United States (US) and Canada, able to provide newly obtained bone marrow aspirate for biomarker analysis.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Female participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment
* Male participants must agree to use a latex condom during sexual contact with females of childbearing potential even if they have had a successful vasectomy starting with the first dose of study treatment through 120 days after the last dose of study treatment
* Able to swallow capsules and able to take or tolerate oral medications on a continuous basis

Dose Determination Arm, Dose Confirmation Arm and Cohort 1 Participants:

* Must have undergone prior treatment with ≥ 2 treatment lines of anti-myeloma therapy and must have failed their last line of treatment
* Prior anti-myeloma treatments must have included an immunomodulatory (IMiD) treatment (lenalidomide, pomalidomide or thalidomide) AND proteasome inhibitor (bortezomib or carfilzomib) alone or in combination and participant must have failed therapy with an IMiD OR proteasome inhibitor
* Must agree to follow the regional requirements for lenalidomide counseling, pregnancy testing, and birth control; willing and able to comply with the regional requirements (for example, periodic pregnancy tests and safety labs)

Cohort 2 Participants:

* MM with relapsing or refractory disease at study entry
* Received prior treatment with 1 to 3 lines for MM
* Achieved a partial response to at least one prior regimen (defined as ≥50% decrease in tumor burden)
* Left ventricular ejection fraction of at least 40%

Exclusion Criteria:

All Participants:

* Currently participating in and receiving study therapy or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study treatment
* History of repeated infections; primary amyloidosis; hyperviscosity; plasma cell leukemia; polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome or Waldenström's macroglobulinemia
* Diagnosis of immunosuppressive disorder or on any other immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Received a prior monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from a baseline AE or a Grade 1 AE associated with agents administered more than 4 weeks earlier
* Prior anti-MM therapy (including dexamethasone), targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or not recovered from AEs due to a previously administered agent
* An additional malignancy that is progressing or requires active treatment within the last 5 years
* Active autoimmune disease or a documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Active infection requiring intravenous systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment
* Prior therapy with an anti-programmed cell death (PD)-1, anti-PD ligand 1 (anti-PD-L1), anti-PD-L2, anti-CD137 antibody, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection
* Clinically significant coagulopathy
* Has had or is planning for allogeneic stem cell transplant
* Autologous stem cell transplant within 12 weeks before the first infusion
* History of Grade 4 rash associated with thalidomide treatment
* Known hypersensitivity to thalidomide, lenalidomide or pomalidomide
* Received a live vaccine within 30 days of planned start of study treatment

Dose Determination Arm, Dose Confirmation Arm and Cohort 1 Participants:

* Clinically active central nervous system (CNS) involvement
* Known gastrointestinal disease that may significantly alter the absorption of lenalidomide
* Unable or unwilling to undergo antithrombotic prophylactic treatment
* Known symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Cohort 2 Participants:

* Smoldering MM (SMM), monoclonal gammopathy of undetermined significance (MGUS), plasma cell leukemia or Waldenström's macroglobulinemia
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to the first dose of study treatment
* Myocardial infarction within 4 months prior to randomization, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless participant has a pacemaker.
* Known history of allergy to CAPTISOL® (a cyclodextrin derivative used to solubilize carfilzomib)
* Hypersensitivity to carfilzomib, bortezomib, boron, or mannitol
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to pre-existing pulmonary or cardiac impairment
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to the first dose of study treatment
* Pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-02-14 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mateos MV, Orlowski RZ, Ocio EM, Rodriguez-Otero P, Reece D, Moreau P, Munshi N, Avigan DE, Siegel DS, Ghori R, Farooqui MZH, Marinello P, San-Miguel J. Pembrolizumab combined with lenalidomide and low-dose dexamethasone for relapsed or refractory multiple myeloma: phase I KEYNOTE-023 study. Br J Haematol. 2019 Sep;186(5):e117-e121. doi: 10.1111/bjh.15946. Epub 2019 May 15. No abstract available. PMID 31090915
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included 3 parts: (1) dose determination/escalation (2) dose confirmation and (3) dose expansion. The study included a pooled analysis of efficacy for participants receiving any dose of pembro+len+dex combined or pembro+carfilzomib (carf)+dex randomized by disease cohort.
Groups:
- Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg: Participants in Part 2 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 200 mg Q2W (Days 1 and 15) in combination with lenalidomide 25 mg (Days 1-21) and dexamethasone 20 mg Q1W during Cycle 1 (28-day cycle).
- Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg: Participants in Part 3 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 200 mg Q2W (Days 1 and 15) in combination with lenalidomide 25 mg (Days 1-21) and dexamethasone 40 mg Q1W during each 28-day cycle.
- Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg: Participants in Part 3 with refractory or relapsed and refractory multiple myeloma (rrMM) received pembrolizumab 200 mg Q2W (Days 1 and 15) in combination with lenalidomide 25 mg (Days 1-21) and dexamethasone 20 mg Q1W during each 28-day cycle.
- Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg: Participants in Part 3 with relapsed or refractory multiple myeloma (rMM) received pembrolizumab 200 mg Q3W in combination with carfilzomib 56 mg/m^2 (Days 1, 2, 8, 9, 15, 16) and dexamethasone 20 mg (Days 1, 2, 8, 9, 15, 16, 22, 23) during each 28-day cycle.
Period: Part 1:Dose Determination/Escalation
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg
Started | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Dose Confirmation
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg
Started | 0 | 0 | 6 (Participants added to study for dose confirmation.) | 2 (Participants added to study for dose confirmation.) | 1 (Participants added to study for dose confirmation.) | 0 | 0 | 0
Treated | 0 | 0 | 6 | 1 | 1 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 6 | 2 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 3:Dose Expansion
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg
Started | 0 | 0 | 0 | 0 | 0 | 47 (Participants added to study for dose expansion) | 1 (Participants added to study for dose expansion) | 10 (Participants added to study for dose expansion)
Treated | 0 | 0 | 0 | 0 | 0 | 45 | 1 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 47 | 1 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2
Not completed — Not Treated | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg | Total
Number analyzed (Participants) | 6 | 4 | 6 | 2 | 1 | 47 | 1 | 10 | 77
Age, Customized [Count of Participants; unit: Participants]
  0 to 17 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 to 64 years | 4 | 2 | 5 | 0 | 0 | 28 | 0 | 8 | 47
  65 to 84 years | 2 | 2 | 1 | 2 | 1 | 19 | 1 | 1 | 29
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 0 | 21 | 1 | 4 | 31
  Male | 5 | 3 | 4 | 1 | 1 | 26 | 0 | 6 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 0 | 0 | 6 | 0 | 2 | 13
  Not Hispanic or Latino | 4 | 1 | 4 | 2 | 1 | 36 | 1 | 2 | 51
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 5 | 0 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 7 | 0 | 0 | 8
  White | 6 | 4 | 5 | 2 | 1 | 39 | 1 | 10 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE v.4.0)
Description: DLTs were assessed during Cycle 1 (28 days) and were defined as the occurrence of any of the following judged by the investigator to be possibly, probably or definitely related to study drug: Grade (Gr) 4 non-hematologic toxicity; Gr 4 hematologic toxicity lasting ≥7 days; Gr 3 non-hematologic toxicity lasting >3 days; Gr 3 non-hematologic laboratory value if: medical intervention was required, abnormality led to hospitalization, was renal or liver function related, or persisted for >1 week; Gr 3/4 febrile neutropenia; thrombocytopenia <25,000 cells/mm^3 (associated with bleeding requiring platelet transfusion or life-threatening bleeding); Gr 5 toxicity; or delay of >1 week in initiating Cycle 2 or unable to complete 80% of treatment during the first course of therapy due to drug-related toxicity. DLTs for the rMM cohort were any drug-related adverse events that cannot be managed by dose modification. DLTs are reported for the maximum tolerated dose.
Time Frame: Up to 28 days in Cycle 1
Population: All DLT-evaluable participants in Parts 1 and 2 who received ≥1 dose of study treatment, completed Cycle 1 (28 days), or who had a DLT during the DLT evaluation period. Per protocol, DLT was not planned to be evaluated in Part 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg
Number analyzed (Participants) | 6 | 3 | 6 | 1 | 1 | 0 | 0 | 0
Participants | 3 | 0 | 0 | 0 | 0 |  |  |

2. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An adverse event was defined as any untoward medical occurrence in a participant administered study treatment and did not necessarily have a causal relationship with this treatment. An adverse event could be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the use of the study treatment was also an adverse event.
Time Frame: Up to approximately 72.7 months
Population: All participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg
Number analyzed (Participants) | 6 | 3 | 6 | 1 | 1 | 45 | 1 | 10
Participants | 6 | 3 | 6 | 1 | 1 | 45 | 1 | 10

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: as for outcome 2
Time Frame: Up to approximately 72.7 months
Population: All participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg
Number analyzed (Participants) | 6 | 3 | 6 | 1 | 1 | 45 | 1 | 10
Participants | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 6

4. Secondary Outcome: Objective Response Rate (ORR) Evaluated According to the International Myeloma Working Group (IMWG) 2006 Response Criteria by Confirmed Investigator Assessment
Description: ORR was the percentage of the participants who achieved at least a partial response (stringent complete response [sCR]+complete response [CR]+very good partial response [VGPR]+partial response [PR]). CR=negative immunofixation of serum and urine+no tissue plasmacytomas+≤5% plasmacytomas in bone marrow; sCR=stringent complete response, CR+normal free light chain (FLC) ratio+no clonal cells in bone marrow; VGPR=serum+urine M-protein detectable by immunofixation but not electrophoresis OR ≥90% reduction in serum M-protein+urine M-protein <100 mg/24 hour(hr); PR = ≥50% reduction of serum M-protein+reduction in 24hr urinary M-protein by ≥90% or to <200 mg/24 hrs.
Time Frame: Up to approximately 72.7 months
Population: The analysis population included all participants who received ≥1 dose of study treatment. The analysis was pre-specified to be a pooled analysis of all participants grouped by disease cohort (rrMM or rMM) and treatment combination (irrespective of dose); therefore data by individual dose were not analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pooled rrMM Cohort: Participants from Parts 1 and 2 with refractory or relapsed and refractory multiple myeloma (rrMM) received any dose combination of pembrolizumab Q2W (Days 1 and 15) in combination with lenalidomide and dexamethasone Q1W during each 28-day cycle.
- Pooled rMM Cohort: Participants from Part 2 with relapsed or refractory multiple myeloma (rMM) received pembrolizumab Q3W in combination with carfilzomib 56 mg/m^2 (Days 1, 2, 8, 9, 15, 16) and dexamethasone 20 mg (Days 1, 2, 8, 9, 15, 16, 22, 23) during each 28-day cycle.
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg | Pooled rrMM Cohort | Pooled rMM Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63 | 10
Percentage of participants |  |  |  |  |  |  |  |  | 30.2 [19.2 to 43.0] | 70.0 [34.8 to 93.3]

5. Secondary Outcome: Disease Control Rate (DCR) Evaluated According to the International Myeloma Working Group (IMWG) 2006 Response Criteria by Confirmed Investigator Assessment
Description: DCR was the percentage of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), or stable disease (SD) ≥12 weeks prior to evidence of disease progression (PD). CR=negative immunofixation of serum and urine+no tissue plasmacytomas+ ≤5% plasmacytomas in bone marrow; sCR=stringent complete response, CR+normal free light chain (FLC) ratio+no clonal cells in bone marrow; VGPR=serum+urine M-protein detectable by immunofixation but not on electrophoresis OR ≥90% reduction in serum M-protein+urine M-protein <100 mg/24 hour(hr); PR=≥50% reduction of serum M-protein+reduction in 24 hr urinary M-protein by ≥90% or to <200 mg/24 hrs; SD=not meeting the criteria for CR, VGPR, PR, or PD. PD=≥1 of the following: ≥25% increase from baseline in serum/urine M-protein; hypercalcemia; increase in FLC ratio; ≥10% bone marrow plasma cells; new or increase in the size of existing bone lesions or tissue plasmacytomas.
Time Frame: Up to approximately 72.7 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg | Pooled rrMM Cohort | Pooled rMM Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63 | 10
Percentage of participants |  |  |  |  |  |  |  |  | 84.1 [72.7 to 92.1] | 100.0 [69.2 to 100.0]

6. Other Pre Specified Outcome: Duration of Response (DOR) Evaluated According to the International Myeloma Working Group (IMWG) 2006 Response Criteria by Confirmed Investigator Assessment
Description: DOR was the time from first evidence of response (stringent complete response [sCR]+complete response [CR], very good partial response [VGPR], partial response [PR]) until disease progression (PD) or death. CR=negative immunofixation of serum and urine+no tissue plasmacytomas+≤5% plasmacytomas in bone marrow; sCR=stringent complete response, CR+normal free light chain (FLC) ratio+no clonal cells in bone marrow; VGPR=serum+urine M-protein detectable by immunofixation but not electrophoresis OR ≥90% reduction in serum M-protein+urine M-protein <100 mg/24 hour(hr); PR = ≥50% reduction of serum M-protein+reduction in 24hr urinary M-protein by ≥90% or to <200 mg/24 hrs. PD=≥1 of the following: ≥25% increase from baseline serum/urine M-protein; hypercalcemia; increase between involved/uninvolved FLC levels; ≥10% bone marrow plasma cells; new or increase in the size of existing bone lesions or tissue plasmacytomas. DOR was calculated using the Kaplan-Meier method for censored data.
Time Frame: Up to approximately 72.7 months
Population: The analysis population included all participants who received ≥1 dose of study treatment and demonstrated at least a partial response. The analysis was pre-specified to be a pooled analysis of all participants grouped by disease cohort (rrMM or rMM) and treatment combination (irrespective of dose); therefore data by individual dose were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg | Pooled rrMM Cohort | Pooled rMM Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 7
Months |  |  |  |  |  |  |  |  | 16.4 [7.7 to 36.8] | 14.1 [8.8 to 17.7]

7. Other Pre Specified Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. OS was calculated from product-limit (Kaplan-Meier) method for censored data. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Time Frame: Up to approximately 72.7 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg | Pooled rrMM Cohort | Pooled rMM Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63 | 10
Months |  |  |  |  |  |  |  |  | 29.0 [17.8 to 42.4] | 22.5 [2.0 to NA] — OS upper limit could not be estimated due to insufficient number of events at the time of final analysis.

8. Other Pre Specified Outcome: Progression Free Survival (PFS) Evaluated According to the International Myeloma Working Group (IMWG) 2006 Response Criteria by Confirmed Investigator Assessment
Description: PFS was defined as the time from randomization to the first documented disease progression (PD) or death due to any cause. PD= ≥1 of the following: ≥25% increase from baseline in serum/urine M-protein; hypercalcemia; increase in FLC ratio; ≥10% bone marrow plasma cells; new or increase in the size of existing bone lesions or tissue plasmacytomas. The median PFS was calculated from the Kaplan-Meier method for censored data.
Time Frame: Up to approximately 72.7 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg | Pooled rrMM Cohort | Pooled rMM Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63 | 10
Months |  |  |  |  |  |  |  |  | 5.6 [2.8 to 7.2] | 14.3 [2.0 to 19.6]

9. Other Pre Specified Outcome: Time to Progression (TTP) Evaluated According to the International Myeloma Working Group (IMWG) 2006 Response Criteria by Confirmed Investigator Assessment
Description: TTP was defined as the time from the first dose to first documented disease progression (PD) or death due to any cause. PD= ≥1 of the following: ≥25% increase from baseline in serum/urine M-protein; hypercalcemia; increase in FLC ratio; ≥10% bone marrow plasma cells; new or increase in the size of existing bone lesions or tissue plasmacytomas.
Time Frame: Up to approximately 72.7 months
Population: All participants who received ≥1 dose of study treatment. The analysis was pre-specified to be a pooled analysis of participants grouped by disease cohort (rrMM or rMM)/treatment (irrespective of dose). There were insufficient data available to conduct the TTP analyses.
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg | Pooled rrMM Cohort | Pooled rMM Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 72.7 months
Description: The analysis population for adverse events (AEs) consisted of all participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE unless considered related to study treatment. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "neoplasm progression", "malignant neoplasm progression" and "disease progression" not related to study treatment are excluded. All-cause mortality is reported for all randomized participants.
Arm/Group | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg
All-Cause Mortality (participants affected / at risk) | 3/6 | 3/4 | 1/6 | 0/2 | 0/1 | 31/47 | 0/1 | 6/10
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/3 | 2/6 | 1/1 | 1/1 | 19/45 | 0/1 | 9/10
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 6/6 | 1/1 | 1/1 | 44/45 | 1/1 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg (N=6) | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg (N=3) | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg (N=6) | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg (N=1) | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg (N=1) | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg (N=45) | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg (N=1) | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 5 (5)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
West Nile viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:Pembro 2mg/kg+Len 25mg+Dex 40 mg (N=6) | Part 1:Pembro 2mg/kg+Len 10 mg+Dex 40 mg (N=3) | Part 2:Pembro 200 mg+Len 25 mg+Dex 40 mg (N=6) | Part 2:Pembro 200 mg+Len 25 mg+Dex 20 mg (N=1) | Part 2:Pembro 200 mg+Len 10 mg+Dex 40 mg (N=1) | Part 3:Pembro 200 mg+Len 25 mg+Dex 40 mg (N=45) | Part 3:Pembro 200 mg+Len 25 mg+Dex 20 mg (N=1) | Part 3:Pembro 200 mg+Carf 56 mg/m^2 +Dex 20 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 17 (32) | 1 (1) | 5 (11)
Neutropenia (Blood and lymphatic system disorders) | 4 (18) | 2 (4) | 2 (16) | 1 (5) | 0 (0) | 17 (45) | 1 (1) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (36) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 18 (38) | 1 (1) | 3 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (5) | 4 (9) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 8 (21) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 2 (2) | 5 (16) | 0 (0) | 1 (6) | 10 (22) | 1 (1) | 4 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 7 (13) | 0 (0) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (12) | 0 (0) | 2 (3)
Asthenia (General disorders) | 1 (4) | 1 (2) | 2 (4) | 1 (1) | 0 (0) | 8 (9) | 0 (0) | 3 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 1 (6) | 11 (29) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 7 (12) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 4 (6)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (3)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tongue fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (11) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 6 (10) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 2 (7)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 2 (13) | 1 (2) | 0 (0) | 9 (15) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 6 (7) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 1 (1) | 8 (9) | 0 (0) | 3 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (10) | 0 (0) | 1 (1) | 7 (23) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (12) | 1 (1) | 1 (2) | 6 (20) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 5 (5) | 0 (0) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 2 (4) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 5 (10) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 10 (14) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (7) | 0 (0) | 0 (0) | 14 (19) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Primary hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid sensory disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment of participants into this study was stopped after the FDA implemented a clinical hold after determining the risks of pembrolizumab + pomalidomide or lenalidomide outweighed any potential benefit for participants with multiple myeloma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT02036502/Prot_SAP_000.pdf